CLINICAL TRIAL: NCT04473612
Title: Degree Physical Status and Upper Airway Function in Neuromuscular Patients
Brief Title: Physical Status and Upper Airway Function in Neuromuscular Patients
Status: Completed | Type: Observational
Sponsor: Universidad de Granada (Other)
Responsible Party: Principal Investigator, Marie Carmen Valenza, Principal Investigator; PT; PhD, Universidad de Granada
Other Study IDs: DF0091UG
Record Dates: First submitted 2020-07-08; First posted 2020-07-16 (Actual); Last update posted 2020-10-14 (Actual); Status verified 2020-10

CONDITIONS: Neuromuscular Diseases; Physical Disability; Airway Disease
MeSH Terms: conditions — Neuromuscular Diseases

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Neuromuscular low physical status group: Patients diagnosed of Neuromuscular disease with low physical status
- Neuromuscular high physical status group: Patients diagnosed of Neuromuscular disease with high physical status
- Control group: Healthy subjects

SUMMARY:
Inside of studies that report an upper airway function impaired, the upper limb strength has been demonstrated to be determinant in breath, speech and swallow performance. Nevertheless, no previous studies in neuromuscular disease have explored the relation between general disability and upper airway function.

There is a suspicion of upper airway which is associated with physical deterioration, however the extent to which if feeds back has not been explored.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of Neuromuscular disease
* Between 6 and 65 years
* Impairment of the upper airway
* Accepted to sign the informed consent

Exclusion Criteria:

* Cognitive impairment.
* Diagnose of autism spectrum disorder or severe intellectual disability
* Physical or functional impairment that limits the performance of evaluation

Ages: 6 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Patients diagnosed of neuromuscular disease aged 6-65 years with an impairment of the upper airway, whether in ventilatory, deglutory or communication capacity.
Sampling Method: Probability Sample
Enrollment: 41 (Actual)
Dates: Start 2020-07-20 (Actual); Primary Completion 2020-08-15 (Actual); Study Completion 2020-09-01 (Actual)

PRIMARY OUTCOMES:
Hand grip strength | Baseline
  Hand grip strength will be evaluated with a pressure dynamometer according to the protocol, to their maximum ability in a seated position . The average of three attempts for the dominant hand will be recorded.
  It has been proven that it can be used as an indicator of general health and as a strong predictor of future mortality, disability, falls, complications and resource utilization.
Respiratory function | Baseline
  Respiratory function will be evaluated with spirometry following standardized protocols. Collected variables will be Forced Expiratory Volume in the First Second (FEV1), Forced Vital Capacity (FVC) and Maximal Voluntary Ventilation (MVV).
Peak expiratory flow | Baseline
  Peak expiratory flow is a person's maximum speed of expiration, as measured with a peak flow meter, a small, hand-held device used to monitor a person's ability to breathe out air. It will be measured following standardized protocols.

SECONDARY OUTCOMES:
European Quality of Life-5 Dimensions (EQ-5D) | Baseline
  The perception of the level of health and the quality of life were evaluated with the questionnaire European Quality of Life-5 Dimensions (EQ-5D). It is composed of 2 parts in which health status is assessed:
  * Descriptive system: It consists on 5 dimensions that include mobility, self-care, usual activities, pain/discomfort, and anxiety/depression. Patients classify their health status in 3 severity levels: having no problems, having some or moderate problems, being unable to do/having extreme problems.
  * Visual Analog Scale, by which respondents can report their perceived health status with a grade ranging from 0 (the worst possible health status) to 100 (the best possible health status).
Fatigue Severity Scale | Baseline
  Fatigue severity scale (FSS) will be used to measure fatigue. It consists of 9 items with answers that the patient scores between 1 and 7. The total is calculated by adding all the items. For children will be used The PedsQL™ Multidimensional Fatigue Scale, which is composed of 18 items comprising 3 dimensions (general fatigue, sleep/rest fatigue, cognitive fatigue), evaluated thorough a Liker scale with values from 0 (never) to 4 (almost always), referring to difficulty presented.
World Health Organization Disability Assessment Scale (WHODAS) 2.0 (WD2) | Baseline
  To measure the degree of disability, the World Health Organization Disability Assessment Scale, WHODAS 2.0 (WD2) will be used. It measures changes in functioning and levels of difficulty in carrying out and carrying out its activities . The WD2 scale is composed of 36 items divided into 6 domains, evaluated through a Likert scale with values from 1 to 5, referring to the difficulty presented. Higher scores show a greater degree of disability.
Activity Limitations in Children and Adults With Neuromuscular Disorders (ACTIVLIM) | Baseline
  The Activity Limitations in Children and Adults With Neuromuscular Disorders (ACTIVLIM) questionnaire is an instrument to measure functional limitation and has been calibrated in children and adults with neuromuscular diseases, according to the difficulty of patients to perform daily activities that require the use of the upper extremities and / or lower.
Brief pain inventory | Baseline
  For pain assessment we will use a specific brief pain questionnaire, Brief Pain Inventory , which consists of three parts. In the first, the patient will indicate in a drawing the area in which he presents this pain. The second part refers to the pain felt in the last days, where it is scored, as in the previous questionnaire, from 0 to 10 (0 being no pain and 10 being the maximum pain felt). Finally, in a third part we see how that pain influences the different activities that the patient performs in his day to day.
Hospital Anxiety and Depression Scale | Baseline
  Anxiety and depression will be assessed with the Hospital Anxiety and Depression Scale (HADS) . This scale is composed of 14 items divided into two subscales, 7 items of anxiety and 7 items of depression, involving higher values worse psycho-emotional state.
Muscle strength of the neck | Baseline
  To evaluate the muscle strength of the neck in neuromuscular patients, neck dynamometry will be performed. With subtests in which front bending, extension, pure lateral flexion, lateral flexion with rotation and pure rotation were measures.
Eating Assessment Tool-10 (EAT-10) | Baseline
  The EAT-10 is a self-administered instrument that evaluate specific symptoms of dysphagia with 10 items and each item have a range from zero (no problem to swallow) to four (a serious problem for life).
  In the case of patients pediatric with dysphagia it used Pediatric Eating Assessment Tool (PEDI-EAT-10)
Swallowing quality of life questionnaire (SWAL-QOL) | Baseline
  To measure the possible swallowing problems in daily life we will used the SWAL-QOL, it contains 44 items and each item was scored from zero (the worst state) to four (the best state) . This questionnaire consists of 44 items, consisting of 11 subscales. With a Likert type score in which the patient scores between 1 and 5. Where 1 indicates the worst state and 5 the most favorable.
Functional Oral Intake Scale (FOIS) questionnaire | Baseline
  The severity of swallowing will be assessed using the Functional Oral Intake Scale (FOIS) questionnaire . This scale consists of 7 levels, with 1 being the most severe and 7 being the least severe, the patient has to select the level with which he is.
Karaduman Chewing Performance Scale (KCPS) | Baseline
  There are also questionnaires like Karaduman Chewing Performance Scale (KCPS) , that permitted us evaluate the function of chewing, this test has not been used in previous studies in adults, so in this study we have only used it in the childrens patients.
Orofacial Myofunctional Evaluation with Scores (OMES) | Baseline
  Clinical evaluation of the orofacial myofunctional condition will be evaluated using the Orofacial Myofunctional Evaluation with Scores (OMES) . It consisting of 4 subscales: appearance and posture, mobility and functions (breathing, deglutition, mastication). The examiner attributed scores on a 3 point scale: 3=normal, 2= insufficient ability; and 1= absence of ability or being unable to perform the task.
Volume Viscosity Clinical Exploration Method (MECV-V) | Baseline
  Volume Viscosity Clinical Exploration Method (MECV-V) , this test provides us with information about the volume to which the 5ml, 10ml and 20 ml patients are able to feed and tells us what viscosity, nectar, liquid and pudding. It is used in the diagnosis of oropharyngeal dysphagia.
Voice handicap index (VHI-30) | Baseline
  The phonatory function and it´s repercussion on daily life will be evaluated by the Voice handicap index (VHI-30) . This scale consists of 30 items, consisting of 3 subscales, functional, physical and emotional. In which the patient must indicate the presence or symptoms of dysphonia with a Likert type score of 5 points, in which 0 indicates never and 4 always indicates.
Grade, Roughness, Breathing, Asthenia, Effort (GRBAS) | Baseline
  Perceptual scale of Grade, Roughness, Breathing, Asthenia, Effort (GRBAS) . Will be used to analyze qualitative aspects of the voice, it is completed by the evaluator who qualifies as: 0 normal, 1 mild, 2 moderate, 3 severe, each quality of the voice (Degree of dysphonia, scratchy, blown, weak or asthenic, tight or strangled).
Functional evaluation of the voice | Baseline
  The functional evaluation of the voice will allow us to measure the intensity, frequency and duration of the voice: To evaluate the intensity of the voice, measured in decibels (dB), we will use a sound level meter; To evaluate the frequency of the voice , measured in Hz (Hz), we use the PRAAT software (Praat from the Dutch "speak"). In addition, the duration of the phonation and breathing times , measured in Sg, will be evaluated, for this we use an audio recorder.

CONTACTS AND LOCATIONS:
Locations (1):
- University of Granada, Granada, Spain

IPD SHARING:
Plan to Share IPD: No